CLINICAL TRIAL: NCT05272267
Title: Transforming ED Throughput With AI-Driven Clinical Decision Support System (TEDAI): The Impact on the Delivery of Care and Patient Experience
Brief Title: Transforming ED Throughput With AI-Driven Clinical Decision Support System
Acronym: TEDAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 202108090RINC
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2022-07

CONDITIONS: Critical Care; Emergency Treatment; Triage; Readmission
Keywords: Critical Care; Emergency Treatment; Triage; Readmission

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted (Active Comparator): AI-assisted models providing diagnosis and prognostic information
  Interventions: Other: AI-assisted models providing diagnosis and prognostic information
- Usual care (Placebo Comparator): usual care without AI-assisted models providing diagnosis and prognostic information
  Interventions: Procedure: Critical treatment

INTERVENTIONS:
Other: AI-assisted models providing diagnosis and prognostic information — AI-assisted models providing diagnosis and prognostic information in the ED, including triage, ICD coding, chest x ray alerts, critical event alerts, readmission prediction, and post-cardiac arrest prognostication.
  Arms: AI-assisted
Procedure: Critical treatment — Critical treatment of the emergency room
  Arms: Usual care

SUMMARY:
The aims of this study is to integrate real-time data flow infrastructure between hospital information system and AI models and to conduct a cluster randomized crossover trial to evaluate the efficacy of the AI models in improving patient flow and relieving ED crowding.

ELIGIBILITY:
Inclusion Criteria:

* ED patients aged 20 years or older
* Patients were treated by the recruited 16 ED attendings.

Exclusion Criteria:

* Patients aged less than 20 years.
* Patients were not treated by the recruited 16 ED attendings.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4016 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
ED length of stay | From ED arrival to 3 days after ED discharge. For hospitalized patients with cardiac arrest, the outcome ascertainment continues until hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Huang, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan